CLINICAL TRIAL: NCT00680719
Title: Preventing HIV/Aids in Tx-Resistant Drug-Abusing Youth
Brief Title: Preventing HIV/Aids in Drug Abusing Youth
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA17023
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: HIV Infections
Keywords: substance abuse; HIV risk; Behavior and Mental Disorders; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders; Behavior; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Family Therapy plus HIV prevention
  Interventions: Behavioral: IBFT /HIV prevention
- 2 (Active Comparator): Family Therapy only.
  Interventions: Behavioral: IBFT

INTERVENTIONS:
Behavioral: IBFT /HIV prevention — Integrated Behavioral and Family Therapy (IBGT) with HIV prevention.
  Arms: 1
Behavioral: IBFT — Integrated Behavioral and Family Therapy (IBFT).
  Arms: 2

SUMMARY:
This project involves two studies focusing on the engagement and treatment of adolescents diagnosed with substance use disorders. Study 1 will evaluate a promising parent-based engagement intervention, Community Reinforcement Training, designed to facilitate the entry of resistant drug-abusing adolescents in treatment. The approach will be compared with an Engagement As Usual intervention condition. Study 2 involves a controlled clinical trial evaluating the efficacy of an HIV/AIDS prevention intervention embedded in family-based drug abuse treatment for reducing HIV/AIDS risk behaviors and substance use. Adolescents who are successfully engaged in treatment through Study 1 will be randomly assigned to receive either family therapy alone or family therapy with the integrated HIV/AIDS prevention intervention. Both studies are being conducted in Portland, Oregon.

ELIGIBILITY:
Inclusion Criteria:

* Parents have an adolescent in the ages of 15-20 years.
* Have had contact with the adolescent on at least 40% of the past 90 days.
* Have some knowledge or evidence that the adolescent would meet DSM-IV diagnostic criteria for a substance abuse disorder.
* Adolescent has explicitly refused to attend any intake or therapy sessions.
* All parents' efforts to enter adolescent into treatment have failed, despite therapist's assistance.
* Residence in Portland vicinity.
* Sufficient residential stability to permit probable contact at follow-up. (e.g. not homeless at time of intake)

Exclusion Criteria:

* Evidence of psychotic or organic state of sufficient severity to interfere with understanding of study instruments and procedures.
* Adolescent has received residential drug treatment longer than a 2-week period in the past 90 days.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 111 (Actual)
Dates: Start 2004-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Changes in adolescent's substance use. | 12 months

SECONDARY OUTCOMES:
Changes in HIV risk behaviors. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Holly B Waldron, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute Center for Family and Adolescent Research, Portland, Oregon, United States